CLINICAL TRIAL: NCT00045279
Title: Phase II Trial of PEG-Intron in Patients With Advanced Renal Cell Carcinoma
Brief Title: PEG-Interferon Alfa-2b in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 01-143; CDR0000256464 (Registry Identifier: PDQ (Physician Data Query)); NCI-G-02-2102
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — peginterferon alfa-2b

INTERVENTIONS:
Biological: PEG-interferon alfa-2b

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may stop the growth of kidney cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of PEG-interferon alfa-2b in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of PEG-interferon alfa-2b in patients with metastatic renal cell carcinoma.
* Determine the time to disease progression in patients treated with this drug.
* Determine the safety of this drug in these patients.
* Determine the quality of life of patients treated with this drug.
* Determine the effect of this drug on biological surrogates of antitumor activity (basic fibroblast growth factor, vascular endothelial growth factor, and interleukin-6 serum levels) in these patients.

OUTLINE: Patients receive PEG-interferon alfa-2b subcutaneously once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at 2 weeks and at 2, 4, 8, and 12 months after initiation of study therapy, and then at completion of study therapy.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Metastatic disease
  * No prior therapy for advanced disease
* Tumor sample available for molecular analysis with prior registration on MSKCC IRB # 89-076
* Bidimensionally measurable disease
* No brain metastases unless completely resected and without evidence of recurrence for at least six months

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2.5 times upper limit of normal (unless due to hepatic metastases)
* Hepatitis B surface antigen negative
* Hepatitis C negative

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* No severe cardiac disease
* No New York Heart Association class III or IV cardiac disease
* No myocardial infarction within the past 12 months
* No ventricular tachyarrhythmias requiring ongoing treatment
* No unstable angina

Pulmonary

* No severe asthma requiring chronic systemic steroids

Other

* HIV negative
* Negative pregnancy test
* Fertile patients must use effective contraception
* No malignancy within the past 2 years except basal cell or squamous cell skin cancer, superficial bladder cancer, or localized prostate cancer

  * Patients who have undergone potentially curative therapy and have been deemed to be at low risk for recurrence are eligible
* No medically significant psychiatric disease (e.g., endogenous depression, psychosis, or bipolar disease) requiring hospitalization
* No prior or active autoimmune disease
* Medically controlled diabetes or thyroid dysfunction allowed
* No clinically significant acute viral or bacterial infection that requires specific therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interleukin-2
* No prior interferon alfa
* No concurrent cytokines or biological response modifiers except epoetin alfa in the case of hematologic compromise
* No concurrent tumor vaccines
* No concurrent monoclonal antibodies
* No concurrent bone marrow/stem cell transplantation

Chemotherapy

* No concurrent cytotoxic agents

Endocrine therapy

* No concurrent high-dose systemic steroids
* Concurrent low-dose corticosteroids (e.g., asthma inhalers, topical creams, or intra-articular injections) allowed
* No concurrent hormonal therapy (including megestrol)
* Concurrent hormone replacement therapy or oral contraceptives allowed

Radiotherapy

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior major surgery
* Concurrent nephrectomy allowed

Other

* At least 14 days since prior anti-infectious therapy
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Feldman DR, Kondagunta GV, Schwartz L, Patil S, Ishill N, DeLuca J, Russo P, Motzer RJ. Phase II trial of pegylated interferon-alpha 2b in patients with advanced renal cell carcinoma. Clin Genitourin Cancer. 2008 Mar;6(1):25-30. doi: 10.3816/cgc.2008.n.004. PMID 18501079
- [Result] Motzer RJ, Rakhit A, Thompson J, Gurney H, Selby P, Figlin R, Negrier S, Ernst S, Siebels M, Ginsberg M, Rittweger K, Hooftman L. Phase II trial of branched peginterferon-alpha 2a (40 kDa) for patients with advanced renal cell carcinoma. Ann Oncol. 2002 Nov;13(11):1799-805. doi: 10.1093/annonc/mdf288. PMID 12419754